CLINICAL TRIAL: NCT05142319
Title: Heterologous Prime-boost-boost Vaccine Combinations for Long-term Humoral and Cellular Immunity Against COVID-19
Brief Title: Efficacy of Different COVID-19 Vaccine Combinations in Inducing Long-term Humoral Immunity [PRIBIVAC]
Acronym: PRIBIVAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: A*Star (Other); KK Women's and Children's Hospital (Other Government); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Barnaby Young, Senior Consultant, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/00821
Record Dates: First submitted 2021-11-30; First posted 2021-12-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
Keywords: Vaccine booster; SARS-CoV-2; Coronavirus; Antibody; Humoral immunity; Cellular immunity; Immunogenicity
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BBV152 COVID-19 vaccine; NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Who Masked: Participant
Masking Description: Only study participants will be blinded to the vaccine allocation. This is to reduce the risk of bias in participant-reported AEs. The study participant will be unblinded at Day-28 visit (Visit 3).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Homologous mRNA booster vaccine (Active Comparator): BNT162b2 + BNT162b2 + BNT162b2 or mRNA-1273 + mRNA-1273 + mRNA-1273
  Interventions: Biological: Homologous mRNA booster vaccine
- Heterologous mRNA booster vaccine (Experimental): BNT162b2 + BNT162b2 + mRNA-1273 or mRNA-1273 + mRNA-1273 + BNT162b2
  Interventions: Biological: Heterologous mRNA booster vaccine
- COVAXIN (Experimental): BNT162b2 + BNT162b2 + COVAXIN or mRNA-1273 + mRNA-1273 + COVAXIN
  Interventions: Biological: COVAXIN
- Nuvaxovid (Experimental): BNT162b2 + BNT162b2 + Nuvaxovid or mRNA-1273 + mRNA-1273 + Nuvaxovid
  Interventions: Biological: Nuvaxovid

INTERVENTIONS:
Biological: Homologous mRNA booster vaccine — Single intradermal injection. The vaccine dose will be according to manufacturer's instructions.
  Arms: Homologous mRNA booster vaccine
Biological: Heterologous mRNA booster vaccine — Single intradermal injection. The vaccine dose will be according to manufacturer's instructions.
  Arms: Heterologous mRNA booster vaccine
Biological: COVAXIN — Single intradermal injection at 6ug (0.5ml) per dose.
  Arms: COVAXIN
Biological: Nuvaxovid — Single intradermal injection at 5mcg (0.5mL) per dose.
  Arms: Nuvaxovid

SUMMARY:
PRIBIVAC will assess a heterologous prime-boost-boost strategy in comparison with a homologous regimen in order to compare short and long-term immunogenicity of different COVID-19 vaccine combinations against the ancestral SARS-CoV-2 as well as different variants of concern (VOCs). Initial phases of the study (Phases A-C) have studied homologous versus heterologous vaccines at the first booster, later phases (Phase D) will study these as the second booster.

Hypothesis: One or more heterologous prime-boost-boost COVID-19 vaccine combinations will produce humoral and cellular immunity that is non-inferior to an homologous prime-boost-boost vaccination against wildtype SARS-CoV-2 and/or 1≥ VOC. In Phases A-C of the study the primary 2 dose mRNA vaccine series was defined as 'Prime-boost'. For phase D we will define these 2 doses as 'Prime' and the 3rd vaccine dose as 'Boost'.

DETAILED DESCRIPTION:
The COVID-19 pandemic has spurred vaccine development and phase 1/2/3 clinical trials in record time. In Singapore, novel mRNA vaccines produced by Pfizer-BioNTech (BNT162b2) and Moderna (mRNA-1273) were the first COVID-19 vaccines to receive interim authorisation under the Pandemic Special Access Route (PSAR). Vaccination in Singapore started first for frontline and healthcare workers with BNT162b2 at the end of December 2020. Over the following months this vaccine program was extended first to older adults and then the general population, while mRNA-1273 was also introduced alongside BNT162b2.

While the pivotal phase 3 clinical trials of BNT162b2 and mRNA-1273 have reported a vaccine efficacy of >95% against symptomatic and severe disease, waning antibody levels and the emergence of variants of concern (VOCs) capable of evading protective immunity (from a wildtype SARS-CoV-2 virus vaccine) have raised the need for a long term COVID-19 immunisation strategy. The emergence of the highly transmissible Omicron VOC in November 2021 heralded a shift in booster vaccination policy in Singapore and overseas. First, recommendations for a third dose of an mRNA vaccine were strengthened and in Singapore receipt of a booster dose within 9 months of completing the primary vaccine series was mandated for maintenance of vaccinated status. Following these efforts booster vaccination uptake increased markedly, and currently 79% of the total population in Singapore has received their first booster vaccination dose. Secondly, recommendations changed to advise that individuals complete the standard vaccination regimen even if they have had prior COVID-19.

Although the original monovalent COVID-19 vaccines have proven effective at preventing death and severe disease, breakthrough infections and reinfections have become more common in the face of an evolving virus. The ever-mutating Omicron virus has resulted in several sublineages such as BA.1, BA.2, BA.4 and BA.5 that have caused surges in COVID-19 cases worldwide. Lab studies consistently suggest that antibodies triggered by vaccines (targeting the ancestral SARS-CoV-2 strain) are less effective at blocking BA.4 and BA.5 than earlier Omicron strains BA.1 and BA.2. This could leave previously infected and/or vaccinated and boosted individuals vulnerable to multiple Omicron infections. Thus, pharmaceutical companies have moved towards developing variant-based vaccines to ensure individuals maintain a high level of protection. On 31 August 2022, the US FDA authorized the bivalent formulations of the Moderna and Pfizer-BioNTech vaccines for use as a single booster dose at least two months following primary or booster vaccination. Since the first detection of the XBB Omicron subvariant in August 2022 in India, it has been detected in more than 17 countries to-date including Singapore, Australia, Bangladesh, Denmark, Japan and the US. To combat the rising COVID-19 infections and reinfections in Singapore, the bivalent Moderna/Spikevax and bivalent Pfizer-BioNTech vaccines were added to the National Vaccination Programme from October 2022.

Third-dose boosters increase humoral and cellular immunity, but the rapid waning of protection against symptomatic infection with VOCs such as Omicron has prompted countries to call for a fourth-dose vaccination program. However, the clinical need, effectiveness and timing of a fourth-dose vaccine booster remain to be assessed.

This study will assess the immunogenicity and safety of heterologous boost COVID-19 vaccine regimens compared with a homologous boost regimen. In the early phases of this study (Phase A to C) volunteers who previously received a homologous primary vaccine series with BNT162b2 (Comirnaty/Pfizer-BioNTech) or mRNA-1273 (Moderna) were enrolled. With robust data now available about the benefits of a first booster dose of the vaccine, phase D of the study will shift to investigating the second booster dose and will simplify eligibility criteria to reflect heterogeneity in vaccinations received among the Singapore population to date, and the high prevalence of COVID-19 infection during the Omicron wave.

In Phases A-C of this study, the booster vaccine for the control group was the homologous mRNA vaccine (e.g. BNT162b2 + BNT162b2 + BNT162b2 or mRNA-1273 + mRNA-1273 + mRNA-1273), while the heterologous vaccine candidates were an alternative COVID-19 vaccine. For individuals randomised to intervention group 1 the mRNA booster vaccine administered was heterologous to the primary series (e.g. BNT162b2 + BNT162b2 + mRNA-1273 or mRNA-1273 + mRNA-1273 + BNT162b2), while for other intervention groups this included vaccines of alternate designs:

Control group: Homologous mRNA booster vaccine Intervention group 1: Heterologous mRNA booster vaccine (Phase A) Intervention group 2: COVAXIN® (Phase B) Intervention group 3: Nuvaxovid (Phase C)

Vaccine candidates in phases A-C entered the study at different time points and participants were randomised at equal probability to the available intervention arms at the time of randomisation. This will reduce the risk of bias (e.g. participant preference for a certain arm) compared with a non-randomised design. While an ideal scenario is to have all the selected vaccines approved prior to the start of recruitment, due to the unknown time of availability of vaccine candidates A, B and C, and the urgency of the current situation, recruitment to the control and intervention group 1 (Phase A) was initiated from 12 Oct 2021. Intervention group 2 (Phase B) was added in January 2022 and discontinued 15 March 2022 per the recommendation from the Data Safety Monitoring Board, who reviewed the trial's preliminary results from the first 10 COVAXIN recipients up to Day 28 post-booster. Recruitment to Intervention group 3 (Phase C) was terminated prior to initiation due to delays in the availability of Nuvaxovid which despite receiving interim authorisation by HSA in February 2022 has only become available for administration in late May 2022.

As of 18 May 2022 uptake of the first booster has increased to 75% of the population - with a sharp increase in uptake from January 2022 following governmental policy changes to the definitions of vaccinated status. A significant proportion of those who have not taken their booster are expected to have either had COVID-19 during the Omicron wave, which severely restricts the ability of the study to continue as initially designed. Related to this, focus is shifting to longer term strategies with a second COVID-19 vaccine booster program beginning for selected individuals in Singapore in March 2022. Phase D of the study will examine this immune response following a second COVID-19 vaccine booster. Study participants will be randomised to receive one of three vaccines in equal proportions: Comirnaty or Cormirnaty Bivalent (Original/Omicron BA.4/5), Moderna/Spikevax or Moderna/Spikevax Bivalent (Original/Omicron BA.1) or Nuvaxovid. For analysis the reference point for determining homologous and heterologous vaccination regimen may include the primary vaccine series or first booster.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent for participation in this study;
2. Aged ≥21years at the time of study enrolment;
3. Received the second dose of BNT162b2 or mRNA-1273 Coronavirus Disease 2019 vaccines at least 6 months prior to enrolment;
4. Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests and other study procedures.

For Phase D inclusion criteria 3 will be amended to 'Received the first booster dose of BNT162b2 or mRNA-1273 Coronavirus Disease 2019 vaccine at least 5 months prior to enrolment'. Only individuals recommended to receive a second booster dose under MOH recommendations will be enrolled.

Exclusion Criteria:

1. Known history of SARS-CoV-2 or SARS-CoV-1 infection;
2. Previously received an investigational coronavirus vaccine;
3. Previously received a SARS-CoV-2 monoclonal antibody;
4. Current or planned simultaneous participation in another interventional study;
5. A history of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a COVID-19 vaccine, or otherwise have a contraindication to one of the available study vaccines per the approved label;
6. Individuals who are immunocompromised (e.g. active leukaemia or lymphoma, generalised malignancy, aplastic anaemia, solid organ transplant, bone marrow transplant, current radiation therapy congenital immunodeficiency, HIV/AIDS with CD4 lymphocyte count < 200 and patients on immunosuppressant medications);
7. Received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids >/= 20 milligram per day of prednisone equivalent). Topical tacrolimus is allowed if not used within 14 days prior to Day 1;
8. Individuals who are pregnant or breast feeding;
9. Chronic illness that, in the opinion of the study team, is at a stage where it might interfere with trial conduct or completion;
10. Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalised involuntarily;
11. Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures in the opinion of the study team;
12. Moderate or severe acute illness/infection (according to study team's judgement) on the day of vaccination, or febrile illness (temperature ≥ 37.5°C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.

For Phase D of the trial exclusion criteria 1 and 4 will no longer apply: exclusion criteria 1 is no longer relevant as it not a consideration in MOH recommendations for COVID-19 booster vaccination, and exclusion criteria 4 because of the broad recommendations from MOH for keeping up to date with COVID-19 boosters.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 anti-spike immunoglobulins | Day 28
  To determine the presence and levels of anti-SARS-COV-2 in human sera

SECONDARY OUTCOMES:
SARS-CoV-2 anti-spike immunoglobulins | Day 1, 7, 180, 360
  To determine the presence and levels of anti-SARS-COV-2 in human sera
Level of SARS-CoV-2 neutralising antibodies | Day 1, 7, 28, 180, 360
  To examine the neutralising capacity of the antibodies in the human sera
Quantitative T-cell responses to spike proteins | Day 1, 7, 28, 180, 360
  Quantitative T-cell responses to the vaccines will be measured using SARS-CoV-2 peptides from spike protein to stimulate the PBMCs isolated from donor's blood.
Solicited local and systemic reaction | Up to 7 days post-vaccination
  The participant will be given a diary to record all the local and general symptoms experienced after receiving the vaccination.
Changes from baseline in laboratory safety measures (Phases A-C only) | Baseline and 7 days post-vaccination
  Blood will be taken from the participant during screening visit prior to vaccination (also known as baseline) for the following clinical labs: a) Full blood count inclusive of differential blood count and platelet count; b) Liver panel including albumin, total bilirubin, ALP and ALT; c) Renal panel including sodium, potassium and creatinine; d) Cardiology panel including creatine kinase and troponin.
  The results of the above clinical tests will be compared with repeat tests at Day 7 post-vaccination.
Unsolicited adverse events (AEs) | 28 days post-vaccination
  Unsolicited AEs will be assessed via the listed study procedures, safety laboratory tests, and participant self-recorded diary.
Serious adverse events (SAEs) and AEs of special interest (eg. myocarditis, pericarditis), medically attended AEs | Up to 360 days post-vaccination
  A serious adverse event or serious adverse drug reaction is any untoward medical occurrence at any dose that:
  * Results in death.
  * Is life-threatening (immediate risk of death).
  * Requires inpatient hospitalization or prolongation of existing hospitalization.
  * Results in persistent or significant disability/incapacity.
  * Results in congenital anomaly/birth defect.
  * Is a Medically important event.

OTHER OUTCOMES:
Vaccine efficacy | Throughout the study
  Surveillance for COVID-19 infections via RT-PCR, Antigen Rapid Test and/or anti-nucleocapsid (N) assay
Residual mRNA vaccine | Day 7
  To determine whether the administered mRNA vaccine (control group and intervention group 1 only) can be detected in the blood. This will be done via qRT-PCR using primers targeting the sequence of the mRNA for SARS-CoV-2 spike protein.

CONTACTS AND LOCATIONS:
Overall Officials: Barnaby Young, A/Prof, Principal Investigator — National Centre for Infectious Diseases
Locations (1):
- National Centre for Infectious Diseases (NCID), Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
All study findings and documents will be regarded as confidential. The investigators and other study personnel must not disclose such information without prior written approval from the PI. Participant confidentiality will be strictly maintained to the extent possible under the law and local hospital policy. Identifiable information will be removed from any published data.

REFERENCES:
- [Background] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Background] Baden LR, El Sahly HM, Essink B, Kotloff K, Frey S, Novak R, Diemert D, Spector SA, Rouphael N, Creech CB, McGettigan J, Khetan S, Segall N, Solis J, Brosz A, Fierro C, Schwartz H, Neuzil K, Corey L, Gilbert P, Janes H, Follmann D, Marovich M, Mascola J, Polakowski L, Ledgerwood J, Graham BS, Bennett H, Pajon R, Knightly C, Leav B, Deng W, Zhou H, Han S, Ivarsson M, Miller J, Zaks T; COVE Study Group. Efficacy and Safety of the mRNA-1273 SARS-CoV-2 Vaccine. N Engl J Med. 2021 Feb 4;384(5):403-416. doi: 10.1056/NEJMoa2035389. Epub 2020 Dec 30. PMID 33378609
- [Derived] Poh XY, Torres-Ruesta A, Yoong T, Wong N, Tan CW, Rouers A, Chavatte JM, Goh YS, Rao S, Chia PY, Ong SWX, Lee TH, Sadarangani SP, Lin RJH, Neo V, Kam IKJ, Huang Y, Hor PX, Loh CY; PRIBIVAC study group; Yeoh AY, Lim DRX, Chia W, Ren EC, Lin RTP, Fong SW, Renia L, Lye DC, Wang LF, Ng LFP, Young BE. Immunogenicity of mRNA vs. BBV152 vaccine boosters against Omicron subvariants: Final results from Phase B of the PRIBIVAC study, a randomized clinical trial. Vaccine. 2024 Nov 14;42(25):126275. doi: 10.1016/j.vaccine.2024.126275. Epub 2024 Sep 5. PMID 39241318
- [Derived] Goh YS, Fong SW, Hor PX, Loh CY, Wang B, Salleh SNM, Ngoh EZX, Lee RTC, Poh XY, Rao S, Chia PY, Ong SWX, Lee TH, Lim C, Teo J, Pada S, Sun LJ, Ong DLS, Somani J, Lee ES, Maurer-Stroh S, Wang CI, Leo YS, Lye DC, Young BE, Ng LFP, Renia L; NCID Study Group; COVID-19 Cohort Study Group. Variant-Specific IgA Protects Against Omicron Infection. J Infect Dis. 2024 Aug 16;230(2):e287-e291. doi: 10.1093/infdis/jiad525. PMID 37996071
- [Derived] Poh XY, Lee IR, Lim C, Teo J, Rao S, Chia PY, Ong SWX, Lee TH, Lin RJH, Ng LFP, Ren EC, Lin RTP, Wang LF, Renia L, Lye DC, Young BE. Evaluation of the safety and immunogenicity of different COVID-19 vaccine combinations in healthy individuals: study protocol for a randomized, subject-blinded, controlled phase 3 trial [PRIBIVAC]. Trials. 2022 Jun 16;23(1):498. doi: 10.1186/s13063-022-06345-2. PMID 35710572
- [Derived] Poh XY, Tan CW, Lee IR, Chavatte JM, Fong SW, Prince T, Hartley C, Yeoh AYY, Rao S, Chia PY, Ong SWX, Lee TH, Sadarangani SP, Lin RJH, Lim C, Teo J, Lim DRX, Chia W, Hiscox JA, Ng LFP, Ren EC, Lin RTP, Renia L, Lye DC, Wang LF, Young BE. Antibody Response of Heterologous vs Homologous Messenger RNA Vaccine Boosters Against the Severe Acute Respiratory Syndrome Coronavirus 2 Omicron Variant: Interim Results from the PRIBIVAC Study, a Randomized Clinical Trial. Clin Infect Dis. 2022 Dec 19;75(12):2088-2096. doi: 10.1093/cid/ciac345. PMID 35543372